CLINICAL TRIAL: NCT06830122
Title: Effects of Lactobacillus Crispatus LCr86 on Bacterial Vaginosis and Ovarian Function in Women: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Lactobacillus Crispatus LCr86 on Bacterial Vaginosis and Ovarian Function in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2025005
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Patients With Bacterial Vaginosis
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Conventional medication (ornidazole vaginal suppositories for 7 days) + 30B CFU/strip/day LCr86 (before meals);
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Conventional medication (ornidazole vaginal suppositories for 7 days) + maltodextrin, one strip/day (before meals);
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study will last 8 weeks and each subject will receive 4 follow-up visits (week 0, week 4, week 8, week 20).
  Arms: Probiotic group
Dietary Supplement: Placebo — The experimental phase of this study will last 8 weeks and each subject will receive 4 follow-up visits (week 0, week 4, week 8, week 20).
  Arms: Placebo group

SUMMARY:
Lactobacillus crispatus LCr86 was selected as a test preparation to observe its clinical efficacy in an intervention trial of combined antibiotic treatment and evaluate its effect on the cure rate, recurrence rate and vaginal flora of patients with bacterial vaginitis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age, history of sexual activity, premenopausal women;
2. Nugent score ≥ 7 for diagnosis of BV;
3. Signed informed consent.

Exclusion Criteria:

1. Mixed vaginitis, such as vulvovaginal candidiasis (VVC), Trichomonas vaginalis (TV) infection, Chlamydia trachomatis (CT) infection, or gonococcal vaginitis;
2. History of systemic organic or psychiatric disease;
3. Planned pregnancy, breastfeeding, or menstruation;
4. Have used any antibiotics within 5 days of disease onset;
5. Long-term use of contraceptives or immunosuppressants;
6. Hypersensitivity or allergy to known components of the study drug.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cure rates for bacterial vaginitis | 8 weeks
  The Nugent score of ≤3 is considered successful in bacterial vaginosis treatment.